CLINICAL TRIAL: NCT06112418
Title: A Randomized Comparison of Cleerly Coronary Artery Disease Stage-Based Care Versus Risk Factor-Based Care for Primary Prevention of Cardiovascular Events
Brief Title: A Randomized Comparison of Stage-Based Care Versus Risk Factor-Based Care for Prevention of Cardiovascular Events
Acronym: TRANSFORM
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cleerly, Inc. (Industry)
Collaborators: CPC Clinical Research (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 202302CPC
Record Dates: First submitted 2023-10-02; First posted 2023-11-01 (Actual); Last update posted 2026-01-23 (Actual); Status verified 2026-01

CONDITIONS: Diabetes Mellitus, Type 2; PreDiabetes; Metabolic Syndrome
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Prediabetic State; Metabolic Syndrome

STUDY DESIGN:
Intervention Model Description: Prospective, randomized, open blinded endpoint (PROBE), event-driven pragmatic trial
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Risk Factor-Based Care (No Intervention): The risk factor-based care group will be managed by their usual care providers, with an initial pre-randomization assessment of current treatment by a centralized cardiology team to optimize care relative to primary prevention guidelines. During the trial, the centralized cardiology team will monitor the provision of medications prescribed and lab values relative to guidelines, and provide feedback and education to site investigators to support optimization. CCTA results will be centrally archived and will remain blinded to the usual care provider until the end of the study.
- Cleerly Stage-Based Care (Experimental): The Cleerly Stage-Based Care group will receive personalized care centrally managed by a remote cardiologist-led team. They will also receive an initial pre-randomization assessment of current treatment by a centralized cardiology team to optimize care relative to primary prevention guidelines. Cleerly CAD Staging System results will be discussed with participants and serve as the basis for standardized algorithm-supported pharmacotherapy & education, which will be intensified if plaque burden has progressed at 24 months.
  Interventions: Device: The Cleerly CAD Staging System

INTERVENTIONS:
Device: The Cleerly CAD Staging System — The Cleerly CAD Staging System is software that utilizes a proprietary algorithm to identify CAD, stage the severity of CAD when present, and generate a prognostic risk score to inform treatment decisions that support CV disease prevention.
  Arms: Cleerly Stage-Based Care

SUMMARY:
TRANSFORM is a prospective, randomized, open blinded endpoint (PROBE), event-driven, pragmatic trial in patients who are at increased risk for atherosclerotic cardiovascular (CV) disease but with no known symptomatic CV disease. The trial tests the hypothesis that a Cleerly Coronary Artery Disease (CAD) Staging System-based care strategy reduces CV events compared with risk factor-based care.

DETAILED DESCRIPTION:
Cardiovascular disease (CVD) persists as the leading cause of morbidity and mortality worldwide at high societal cost. The current primary CVD prevention strategy relies upon risk stratification using population health markers such as age, sex, diabetes, hypertension, dyslipidemia and tobacco use, with preventive therapy intensified in higher risk strata. Since these risk factors are indirect surrogate markers of the underlying disease, atherosclerosis, this strategy leads to treatment of individuals with risk factors who do not have atherosclerosis and failure to treat those with significant atherosclerosis who lack risk factors. The current strategy also cannot determine which individuals are inadequately treated despite effective risk factor management (residual risk). With the current approach, the CV death rate is trending upward in the US despite evidence that screening asymptomatic patients reduces CV events and the widespread availability of effective preventive therapies.

This randomized, controlled, pragmatic trial is designed to address the unmet need for better strategies to identify asymptomatic individuals at increased risk for CV events due to atherosclerosis and to personalize their treatment based on CV risk estimates using coronary artery disease (CAD) visualization and quantification.

This study enrolls patients without known symptoms of ASCVD but who are at increased risk for ASCVD due to their age and having diabetes, prediabetes or metabolic syndrome and tests the hypothesis that a CAD Staging System-based care strategy reduces CV events compared with risk factor-based care. The Cleerly CAD Staging System incorporates imaging-based evaluation for coronary atherosclerosis, algorithm-supported pharmacotherapy and personalized education about their CAD.

ELIGIBILITY:
Inclusion Criteria:

1. Provided electronic or written informed consent
2. Men > 55, women > 65 years of age
3. Type 2 diabetes mellitus requiring pharmacologic therapy, prediabetes (most recent HbA1c 5.7 to 6.4% and/or fasting glucose 100-125 mg/dL [5.6-6.9 mmol/L]) and/or metabolic syndrome. Metabolic syndrome is defined as > 3 of the following criteria (International Diabetes Federation 2006):

   * Body mass index ≥ 27 kg/m2 or abnormal waist circumference defined as ≥ 80 cm (31.5 inches) for women, ≥ 94 cm (37 inches) for men; for South and East Asian men (e.g., Asian Indian, Chinese, Japanese) ≥ 90 cm (35.4 inches)
   * Fasting triglycerides ≥ 150 mg/dL (1.7 mmol/L) or treated hypertriglyceridemia
   * HDL-cholesterol (HDL-C) < 40 mg/dL (1.03 mmol/L) in men, <50 mg/dL (1.29 mmol/L) in women or treatment for this lipid abnormality
   * Systolic blood pressure (BP) ≥ 130 and/or diastolic BP≥ 85 mm Hg and/or treated hypertension
   * Fasting blood glucose ≥ 100 mg/dL (5.6 mmol/L) or HbA1c ≥ 5.7%
4. Have a device (e.g., smartphone, tablet, computer) for communication with the central cardiologist-led team managing drug treatment for the personalized care group

Exclusion Criteria:

1. History of symptomatic CVD defined as prior MI, exertional or unstable angina, ischemic stroke, claudication, arterial revascularization for atherosclerosis or other CVD being actively managed by a cardiologist, e.g. atrial fibrillation, heart failure
2. Planned arterial revascularization
3. Inability to complete screening CCTA or any condition that would increase the risk associated with CCTA or increase likelihood of uninterpretable scan including:

   1. eGFR < 60 mL/min/1.73 m2 by the Chronic Kidney Disease Epidemiology Collaboration (CKD EPI) or Modification of Diet in Renal Disease (MDRD) equation (www.kidney.org/professionals/kdoqi/gfr_calculator)
   2. Allergy to iodinated contrast or history of contrast-induced nephropathy (including adverse reaction to contrast at screening CCTA) or screening laboratory values consistent with untreated hyperthyroidism. Participants with elevated thyroid-stimulating hormone (TSH) may be enrolled but should be referred to their physician for evaluation for treatment.
   3. Thyroid cancer in the previous five (5) years or planned radioactive iodine treatment
   4. Weight > 300 lbs. (136 kg) or above manufacturer-recommended limit for scanner and table at the site
   5. Inability to hold breath for > 10 seconds
   6. Active arrhythmia (atrial fibrillation, atrial flutter, frequent premature atrial, or ventricular contractions) with poorly controlled rate (i.e., > 80 beats per minute at screening or prior to CCTA)
   7. Contraindication to dosing with beta blocker or nitroglycerin on day of screening CCTA
   8. Any other factor that, in the opinion of the investigator, would increase participant risk or increase the chance of an uninterpretable CCTA
4. Unsuitable as a trial participant in the opinion of the investigator for reasons including significant left main stenosis (e.g. ≥ 70%; site will be notified by Cleerly), other health condition with life expectancy < 3 years or being at risk of poor compliance with study procedures (e.g., active substance abuse or untreated mental illness that, in the opinion of the investigator, is likely to adversely affect adherence or retention)

Min Age: 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 7500 (Estimated)
Dates: Start 2024-03-06 (Actual); Primary Completion 2029-03-05 (Estimated); Study Completion 2029-03-05 (Estimated)

PRIMARY OUTCOMES:
The primary objective is to compare Cleerly stage-based care with risk factor-based care on the risk of CV events. | Through study completion- an average of 3.5 years
  The primary endpoint is total (first and subsequent) events for the composite endpoint of CV death, myocardial infarction (MI), ischemic stroke, acute limb ischemia, clinically driven arterial revascularization, and hospitalization or urgent visit for heart failure.

SECONDARY OUTCOMES:
The secondary objective is to compare Cleerly CAD stage-based care with risk factor-based care on other clinical events of CV and renal morbidity and mortality. | Through study completion- an average of 3.5 years
  The secondary endpoints are time from randomization to first occurence of an event in the primary efficacy endpoint.
The secondary objective is to compare Cleerly CAD stage-based care with risk factor-based care on other clinical events of CV and renal morbidity and mortality. | Through study completion- an average of 3.5 years
  The secondary endpoints are total occurences after randomization of the primary efficacy endpoing, kidney failure, sustained estimated glomerular filtration rate (eGFR) decrease >40% from baseline, and death from renal causes.
The secondary objective is to compare Cleerly CAD stage-based care with risk factor-based care on other clinical events of CV and renal morbidity and mortality. | Through study completion- an average of 3.5 years
  The secondary endpoints are first and total occurrences after randomization of coronary death, MI, and urgent coronary revascularization.
The secondary objective is to compare Cleerly CAD stage-based care with risk factor-based care on other clinical events of CV and renal morbidity and mortality. | Through study completion- an average of 3.5 years
  The secondary endpoints are time from randomization to first occurrence of MI or ischemic stroke.
The secondary objective is to compare Cleerly CAD stage-based care with risk factor-based care on other clinical events of CV and renal morbidity and mortality. | Through study completion- an average of 3.5 years
  The secondary endpoints are time from randomization to all-cause death.

OTHER OUTCOMES:
The safety objective is to assess harm with the 2 prevention strategies | Through study completion- an average of 3.5 years
  The safety endpoints are Adverse events (AE) leading to discontinuation of study-recommended medication (DAE), serious AE (SAE), adverse device effect (ADE).
The safety objective is to assess harm with the 2 prevention strategies | Through study completion- an average of 3.5 years
  The safety endpoints are 20-item Short Form survey (SF-20).

CONTACTS AND LOCATIONS:
Overall Officials: Deepak Bhatt, MD, MPH, Study Chair — Mt. Sinai Heart
Locations (112):
- United States (112):
  - Chandler Clinical Trials, Chandler, Arizona
  - Scottsdale Clinical Trials, Scottsdale, Arizona
  - Sun City Research, Sun City, Arizona
  - Noble Clinical Research, Tucson, Arizona
  - Cardiovascular Research Foundation of Southern California, Beverly Hills, California
  - Amicis Research: Beverly Hills, Beverly Hills, California
  - Valiance Clinical Research - Canoga Park, Canoga Park, California
  - Cardiovascular Institute of San Diego, Chula Vista, California
  - Amicis Research: Granada Hills, Granada Hills, California
  - Valiance Clinical Research: Huntington Park, Huntington Park, California
  - HALO Diagnostics, Indian Wells, California
  - Chemidox Clinical Trials, Lancaster, California
  - Long Beach Research Institute, Long Beach, California
  - Ace Research Institute - Monterey Park, Monterey Park, California
  - Amicis Research: Newhall, Newhall, California
  - Ace Research Institute: Northridge, Northridge, California
  - Amicis Research: Northridge, Northridge, California
  - Ace Research Institute: Northridge #2, Northridge, California
  - Northridge Clinical Trials, Northridge, California
  - Stanford Health Care, Palo Alto, California
  - VA Palo Alto, Palo Alto, California
  - Amicis Research: San Fernando, San Fernando, California
  - Valiance Clinical Research - Tarzana, Tarzana, California
  - Lundquist Institute for Biomedical Innovation at Harbor - UCLA Medical Center, Torrance, California
  - Amicis Research: Valencia, Valencia, California
  - Concierge Clinical Trials, Valley Village, California
  - University of Colorado, Aurora, Colorado
  - St. Josephs (Intermountain Healthcare), Denver, Colorado
  - Flourish Medical Research, Boca Raton, Florida
  - Apex Research, Cross City, Florida
  - Evolution Research Center, Hialeah, Florida
  - UF Health Jacksonville, Jacksonville, Florida
  - Fiel Wellness Clinical Research LLC, Miami, Florida
  - BioPhase Research, Miami, Florida
  - United Clinical Research, Miami, Florida
  - Atlantis Clinical Research, LLC, Miami, Florida
  - Baptist Health Miami Cardiac and Vascular Institute, Miami, Florida
  - Farma Medical Inc., Miami, Florida
  - New Access Research and Medical Center, Miami, Florida
  - Quantum Clinical Trials, Miami Beach, Florida
  - Ascension Sacred Heart, Pensacola, Florida
  - Clinical Research Center of Florida, Pompano Beach, Florida
  - University of South Florida, Tampa, Florida
  - Aiyan Diabetes Center, Augusta, Georgia
  - Emory University, Dunwoody, Georgia
  - Peachtree Clinical Solutions - Noir Research Collective, Powder Springs, Georgia
  - Randomize Now, LLC - Noir Research Collective, Riverdale, Georgia
  - Privia Medical Group Georgia, LLC (Javara Inc.), Savannah, Georgia
  - Privia Medical Group Georgia - Thomasville (Javara), Thomasville, Georgia
  - Care Institute- High Desert, Meridian, Idaho
  - Northshore University Health System, Evanston, Illinois
  - Indiana Medical Research Institute, Indianapolis, Indiana
  - Franciscan Physician Network- Indiana Heart Physicians, Indianapolis, Indiana
  - MercyOne Iowa Heart Center, West Des Moines, Iowa
  - St Elizabeth Health Care - CRI, Edgewood, Kentucky
  - UofL Health, Louisville, Kentucky
  - Flourish Bowie dba Flourish Research, Bowie, Maryland
  - Massachusetts General Hospital, Boston, Massachusetts
  - Brigham and Women's Hospital, Boston, Massachusetts
  - Henry Ford Hospital, Detroit, Michigan
  - Trinity Health Michigan Heart, Ypsilanti, Michigan
  - Minneapolis Heart Institute Foundation, Minneapolis, Minnesota
  - Washington University School of Medicine, St Louis, Missouri
  - Saint Louis Heart and Vascular, St Louis, Missouri
  - Boeson Research Kalispell, Kalispell, Montana
  - Boeson Research Fort Missoula, Missoula, Montana
  - Bryan Heart, Lincoln, Nebraska
  - Southwest Medical Associates- Optum Nevada, Las Vegas, Nevada
  - Vector Clinical Trials, Las Vegas, Nevada
  - Advanced Heart and Vascular Institute of Hunterdon, Flemington, New Jersey
  - Virtua Health, Inc., Marlton, New Jersey
  - Rutgers State University, New Brunswick, New Jersey
  - The Valley Hospital, Paramus, New Jersey
  - Holy Name Medical Center, Teaneck, New Jersey
  - Clindove Research, Brooklyn, New York
  - Swift Clinical Research, Brooklyn, New York
  - Rasaj Research, Jackson Heights, New York
  - Optum- Long Island NY, Lake Success, New York
  - Northwell Health Northern Westchester Hospital, Mount Kisco, New York
  - Mount Sinai West, New York, New York
  - Mount Sinai, New York, New York
  - University of North Carolina at Chapel Hill, Chapel Hill, North Carolina
  - Duke University Hospital, Durham, North Carolina
  - Durham Veterans Affairs Medical Center (Durham VAMC), Durham, North Carolina
  - Cape Fear Valley Health System (Javara Inc.), Fayetteville, North Carolina
  - West Clinical Research, Morehead City, North Carolina
  - Wake Forest University Health Sciences, Winston-Salem, North Carolina
  - Sanford Health, Fargo, North Dakota
  - Summa Health, Akron, Ohio
  - Hightower Clinical, Oklahoma City, Oklahoma
  - Medical Research International, LLC, Oklahoma City, Oklahoma
  - Ascension St. John - Jane Phillips Medical Center, Tulsa, Oklahoma
  - Capital Area Research, Camp Hill, Pennsylvania
  - Medical University of South Carolina, Charleston, South Carolina
  - Community DPC, Cleveland, Tennessee
  - University of Tennessee Medical Center, Knoxville, Tennessee
  - TriStar Centennial Medical Center (HCA Health Care), Nashville, Tennessee
  - Hendrick Health, Abilene, Texas
  - Gadolin Research, Beaumont, Texas
  - CardioVoyage, LLC, Greenville, Texas
  - Helium Research Group, Houston, Texas
  - Kelsey Research Foundation, Houston, Texas
  - The Methodist Hospital, DeBakey Cardiology Associates, Houston, Texas
  - Gulf Coast Clinical Research, LLC, Houston, Texas
  - Aeres Clinical Research, Laredo, Texas
  - DC Clinical Research, Lewisville, Texas
  - North Dallas Research Associates - Kerlo Network, McKinney, Texas
  - SMS Clinical Research, Mesquite, Texas
  - Privia Medical Group Gulf Coast, PLLC ( Javara Inc.), San Marcos, Texas
  - Privia Medical Group- North Texas, Stephenville, Texas
  - Chippenham Johnston Willis Medical Center, Richmond, Virginia
  - Charleston Area Medical Center, Charleston, West Virginia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Tsao CW, Aday AW, Almarzooq ZI, Alonso A, Beaton AZ, Bittencourt MS, Boehme AK, Buxton AE, Carson AP, Commodore-Mensah Y, Elkind MSV, Evenson KR, Eze-Nliam C, Ferguson JF, Generoso G, Ho JE, Kalani R, Khan SS, Kissela BM, Knutson KL, Levine DA, Lewis TT, Liu J, Loop MS, Ma J, Mussolino ME, Navaneethan SD, Perak AM, Poudel R, Rezk-Hanna M, Roth GA, Schroeder EB, Shah SH, Thacker EL, VanWagner LB, Virani SS, Voecks JH, Wang NY, Yaffe K, Martin SS. Heart Disease and Stroke Statistics-2022 Update: A Report From the American Heart Association. Circulation. 2022 Feb 22;145(8):e153-e639. doi: 10.1161/CIR.0000000000001052. Epub 2022 Jan 26. PMID 35078371
- [Background] Clerc OF, Fuchs TA, Stehli J, Benz DC, Grani C, Messerli M, Giannopoulos AA, Buechel RR, Luscher TF, Pazhenkottil AP, Kaufmann PA, Gaemperli O. Non-invasive screening for coronary artery disease in asymptomatic diabetic patients: a systematic review and meta-analysis of randomised controlled trials. Eur Heart J Cardiovasc Imaging. 2018 Aug 1;19(8):838-846. doi: 10.1093/ehjci/jey014. PMID 29452348
- See also: World Health Organization - Cardiovascular Diseases — http://www.who.int/health-topics/cardiovascular-diseases#tab=tab_1